CLINICAL TRIAL: NCT00005361
Title: Determinants of Respiratory Health in Young Adults
Status: Completed | Type: Observational
Sponsor: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Other Study IDs: 4248; R01HL048619 (NIH)
Record Dates: First submitted 2000-05-25; First posted 2000-05-26 (Estimated); Last update posted 2016-05-13 (Estimated); Status verified 2000-06

CONDITIONS: Lung Diseases
MeSH Terms: conditions — Lung Diseases

SUMMARY:
To measure lung function and respiratory symptom status in a large cohort of healthy, non-smoking 18-22 year old subjects, and relate these measurements to past histories of passive smoke and air pollution exposures.

DETAILED DESCRIPTION:
BACKGROUND:

While the natural history of human lung function growth and decline has been studied intensively over the past 30 years, relatively few data have been collected during the period in which peak volumetric function is achieved, i.e., around the age of 20. As a result, very little is known about the factors, both demographic and environmental, which influence maximal attained lung function.

DESIGN NARRATIVE:

The longitudinal study collected information on the history of respiratory illness, residential history, parental smoking, socio-economic status and home characteristics via an initial questionnaire administered to cadets enrolling at West Point. A sequence of four annual measurements of lung function (by spirometry), and prior-year respiratory health status and activity patterns was obtained in the spring of each year. Pollution exposures were estimated by matching residential histories with historical pollution data stored at the Environmental Protection Agency. Data on meteorological variables (temperature, relative humidity, wind speed) and altitude were obtained for each residential location. The four annual lung function measurements provided precise estimates of individual mean levels of FVC, FEV1, FEF25-75, PEFR, and flow rates at 50 percent and 75 percent of expired FVC. Subject-specific lung function level was analyzed in relation to history of parental smoking and prior exposure to air pollution using analysis of variance methods, controlling for potential confounding variables. In addition to testing these hypotheses regarding the respiratory effects of passive smoking and air pollution exposure, the study also explored the effects of these exposures on the change in lung function between the ages of 18 and 22 and on respiratory illness and symptom experience while at West Point. Finally, the study established a cohort which could be followed in future years.

The study completion date listed in this record was obtained from the "End Date" entered in the Protocol Registration and Results System (PRS) record.

ELIGIBILITY:
No eligibility criteria

Max Age: 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Dates: Start 1993-04; Study Completion 1998-03 (Actual)

REFERENCES:
- [Background] Kinney PL, Nilsen DM, Lippmann M, Brescia M, Gordon T, McGovern T, El-Fawal H, Devlin RB, Rom WN. Biomarkers of lung inflammation in recreational joggers exposed to ozone. Am J Respir Crit Care Med. 1996 Nov;154(5):1430-5. doi: 10.1164/ajrccm.154.5.8912760.